CLINICAL TRIAL: NCT07314281
Title: "Comparing Efficacy of Intravenous Azithromycin and Meropenem for Extensively Drug-Resistant Enteric Fever: A Randomized Controlled Trial" (Pilot Study)
Brief Title: Meropenem vs Azithromycin Efficacy in Case XDR Enteric Fever
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Indus Hospital and Health Network (Other)
Responsible Party: Principal Investigator, Muhammad Hamid Hanif, Principal Investigator, Indus Hospital and Health Network
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IHHN_IRB_2024_10_010
Record Dates: First submitted 2025-09-17; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Enteric Fever
MeSH Terms: conditions — Typhoid Fever | interventions — Azithromycin; Meropenem

STUDY DESIGN:
Intervention Model Description: randomized, controlled, parallel open-label pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Meropenem arm (Active Comparator): For the standard care protocol, patients are initially treated with meropenem 1g intravenously every 8 hours. Once their condition stabilizes , treatment is transitioned to oral azithromycin. The transition involves administering a first dose of azithromycin 1g orally, followed by a daily dose of 500mg orally. Intravenous meropenem will continue until 24 hours after the patient's fever has resolved, after which the treatment will switch to oral azithromycin.
  Interventions: Drug: Meropenem Injection
- Azithromycin arm (Experimental): In the intervention group, patients begin with azithromycin 1g administered intravenously for the initial dose, followed by a daily dose of 500mg intravenously. When the patient's condition stabilizes, the treatment will transition to oral azithromycin, starting with a 1g oral dose and continuing with 500mg orally once daily. Intravenous azithromycin will be maintained until 24 hours after the patient's fever has resolved, after which the treatment will switch to oral azithromycin
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Azithromycin — Azithromycin 1g IV loading dose then 500mg IV OD
  Other Names: Experimental group
  Arms: Azithromycin arm
Drug: Meropenem Injection — Meropenem 1000 mg IV Q8H
  Arms: Meropenem arm

SUMMARY:
1. Primary Objective:

   o To evaluate the efficacy of intravenous azithromycin compared with meropenem in the treatment of extensively drug-resistant (XDR) enteric fever.
2. Secondary Objectives:

   * To evaluate the fever defervescence and Salmonella Typhi eradication
   * To evaluate the cost-effectiveness of intravenous azithromycin versus meropenem in treating XDR enteric fever.
3. Exploratory Objectives:

   * To evaluate the drug resistance against intravenous azithromycin versus in treating XDR enteric fever.

DETAILED DESCRIPTION:
Screening Period:

Patients with positive blood culture of XDR S. typhi underwent further screening for inclusion in study by physician. Before randomization, ECG monitoring, investigations including serum creatinine, liver function test, pregnancy test for married female participants will be done. If patient meet eligibility criteria and physician enrolled, randomization will be done and treatment will be allocated.

Treatment Period:

During treatment period, on D3 clearance blood culture will be sent to check bacterial eradication or sterility of blood. Temperature, blood pressure, pulse will be monitored three times a day. If D3 blood culture and sensitivity report is still positive, second clearance blood culture will be sent on D7. On D7 ECG and LFTs will reassessed. On D7 of treatment detailed clinical assessment will be done in order to evaluate improvement in clinical condition and need of therapy modification "Discontinuation of treatment" based on the list of all terms and condition including hypersensitivity reaction, any adverse event. Total treatment duration will be 14 days. Resolution of symptoms, fever defervescence and blood culture clearance will be consider as study end point.

Randomization and Blinding:

The participant meeting all the inclusion and exhibits no characteristics of exclusion criteria will be eligible to enroll in the study. The written informed consent will be taken and signed ICF will be obtained from participant. The participants will be enrolled in the study based on randomization. The randomization will be done by using randomization allocation software. The office of research and innovation (ORIC) personnel independent from the study will randomize and allocate treatment group. This is an open-label study; thus, both the investigators and participants will be aware of the treatment allocation after randomization. Principle investigator will enroll participants in collaboration with physician. The office of research and innovation (ORIC) personnel will develop envelope containing allocation sequence and treatment option either standard treatment or intervention treatment. Envelop will hand over to physician and will assign treatment option to participants.

Study treatment and Intervention:

For the standard care protocol, patients are initially treated with meropenem 1g intravenously every 8 hours. Once their condition stabilizes , treatment is transitioned to oral azithromycin. The transition involves administering a first dose of azithromycin 1g orally, followed by a daily dose of 500mg orally. Intravenous meropenem will continue until 24 hours after the patient's fever has resolved, after which the treatment will switch to oral azithromycin.

In the intervention group, patients begin with azithromycin 1g administered intravenously for the initial dose, followed by a daily dose of 500mg intravenously. When the patient's condition stabilizes, the treatment will transition to oral azithromycin, starting with a 1g oral dose and continuing with 500mg orally once daily. Intravenous azithromycin will be maintained until 24 hours after the patient's fever has resolved, after which the treatment will switch to oral azithromycin.

ELIGIBILITY:
Inclusion Criteria:

* Participants will enrolled on following criteria

  * Voluntarily sign the written informed consent
  * Patient's of age 1-70 years with clinically suspected on physician decision or XDR enteric fever confirmed by blood culture and sensitivity tests.
  * Married females with negative pregnancy test.
  * No history of cardiac issues with ECG abnormalities, cholestatic jaundice/hepatic dysfunction associated with prior azithromycin use.
  * Patients having no hypersensitivity (skin rashes, anaphylaxis) to azithromycin and meropenem
  * Patients on concomitant medication, having no drug-drug interaction with meropenem and azithromycin will be included in study.

Exclusion Criteria:

* Participants will excluded on following criteria

  * Pregnant, lactating women or women of childbearing age with positive pregnancy test at baseline.
  * Patients with known hypersensitivity (skin rashes, anaphylaxis) to azithromycin, meropenem, or any other macrolide or carbapenem antibiotics.
  * Blood culture and sensitivity tests reported positive culture with MDR S. typhi (non-susceptibility to at least one agent in three or more antimicrobial categories,) o
  * Patients with history of cardiac disorder with ECG abnormalities and history of cholestatic jaundice/hepatic dysfunction associated with prior azithromycin use will be excluded.
  * Patients on continuous medication, having drug-drug interaction with meropenem and azithromycin will be excluded.

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Fever defervescence | Mid-treatment outcome (Day 7)
  Proportion of participants with fever defervescence of temperature 37 ℃ at Mid-treatment outcome (Day 7). Temperature will be monitored and documented in degrees centigrade (°C)
Salmonella Typhi eradication | Mid-treatment outcome (Day 7)
  Proportion of participants with Salmonella Typhi eradication in Blood culture test on day 3. After start of intervention, a clearance of blood culture will be monitor at day 3. if Salmonella Typhi in blood culture of day 3 will not eradicate, a second blood culture will be done on Day 7.

SECONDARY OUTCOMES:
Hospital Admission Days | End-of-treatment outcome (Day 14)
  Mean hospital length of stay (in days) will be compared between groups to evaluate differences in duration of hospitalization
Cumulative Treatment Duration | End-of-treatment outcome (Day 14)
  Average total treatment duration, expressed in number of days, will be compared across groups to assess differences in cumulative therapy requirements
Adverse Events Monitoring | Mid-treatment outcome (Day 7)
  Adverse events will be monitored throughout the study period, including abnormal clinical findings such as rash, pruritus, flushing, or angioedema of the face or extremities. Laboratory assessments (ECG and liver function tests) will be performed on Mid-treatment outcome (Day 7) to check any ECG changes and hepatotoxicity. Vital signs-including body temperature (°C), blood pressure (mmHg), and heart rate (beats/min) will be recorded daily from baseline (Day 1) to day of discharge from hospital.
Antimicrobial Resistance and Cost of treatment | End-of-treatment outcome (Day 14)
  Antimicrobial resistance will be assessed by monitoring any changes in the susceptibility pattern of Salmonella Typhi isolates during the study period. The direct cost of treatment will be calculated in Pakistani Rupees (PKR), based on the total cost of vials utilized throughout the treatment course, and will be compared between study groups to evaluate overall cost-effectiveness.

CONTACTS AND LOCATIONS:
Overall Officials: muhammad hamid, Principal Investigator — Indus Hospital and Health Network
Locations (1):
- Indus Hospital & Health Network - Mian Campus, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
will be shared till December 2025